CLINICAL TRIAL: NCT03397056
Title: How Participants Perceive Biomedical Research in Pulmonology
Acronym: PROTOACCEPT2
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0447
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-03

CONDITIONS: Biomedical Research
Keywords: Patient willingness; Participation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: The target population corresponds to patients with a respiratory disease already included in a biomedical research protocol.
  Intervention: Questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The Questionnaire is provided in the links at the end of the declaration.

SUMMARY:
The primary objective of this study is to determine how biomedical research is perceived by patients already participating in a pulmonology research project.

DETAILED DESCRIPTION:
Over time, clinical research has become a challenge both in terms of public health and in terms of scientific progress. Additionally, it has also become a financial challenge for institutions, especially in France where a significant part of their government funding is provided according to their ability to conduct quality clinical research. Pulmonology is a sector where clinical research is well established with strong incentives from several pharmaceutical companies and numerous academic research projects. Nevertheless, it is important to put the patient back at the centre of biomedical research.

A better knowledge of patient expectations, questions and misunderstandings would considerably improve treatment observance, clinical trial data quality, doctor-patient trust/relationship, and ultimately, the patient's health.

The primary objective of this study is to determine how biomedical research is perceived by patients already participating in a pulmonology research project.

The secondary objectives are to determine:

* how biomedical research is experienced / felt;
* if the information delivered to the patient (orally - information note) is clearly perceived.

Comparisons with PROTOACCEPT1 (osf.io/nsjjr) will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* The patient presents with at least one of the following: (1) asthma, (2) chronic obstructive pulmonary disease, (3) bronchiectasis, (4) idiopathic pulmonary fibrosis, (5) pulmonary arterial hypertension, (6) sleep apnoea syndrome
* The patient is participating in a biomedical research protocol.

Exclusion Criteria:

* Patient under 18 years of age
* Patient judged incapable of filling out the questionnaire for linguistic or other reasons.
* The patient has already participated in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population corresponds to patients with a respiratory disease already included in a biomedical research protocol.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The PROTOACCEPT2 questionnaire. | day 0 (transversal study)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD, PhD, Study Director — University Hospitals of Montpellier
Locations (2):
- France (2):
  - APHM - Hôpital Nord, Marseille
  - CHRU Montpellier - Hôpital Arnaud de Villeneuve, Montpellier

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study. Data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  Data will be made available on a not-for-profit, free platform that allows access control: zenodo.
  A link on osf.io/pxnhc will point towards the zenodo upload.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Individual datasets will be made available at time of submission.
Access Criteria: The conditions under which members of the public will be granted access to the uploaded files are:
  * The user does not work for a private insurance company;
  * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a patient or group of patients;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.
URL: http://osf.io/pxnhc

REFERENCES:
- See also: PROTOACCEPT2 on the Open Science Framework (access to questionnaire) — http://osf.io/pxnhc